CLINICAL TRIAL: NCT01711619
Title: Interventional, Prospective, Multicenter, Randomized, Parallel-arm Study to Compare the Effectiveness of Peripheral Nerve Stimulation (PNS) Utilizing a Subcutaneous Lead Implant Technique (SQS) Plus Optimized Medical Management (OMM) Versus OMM Alone in Patients Suffering From Back Pain Due to Failed Back Surgery Syndrome (FBSS)
Brief Title: SubQStim: A Post-market Study of Subcutaneous Nerve Stimulation in Failed Back Surgery Syndrome (FBSS) Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Challenges to recruit qualified participants
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1.02.7007
Record Dates: First submitted 2012-07-12; First posted 2012-10-22 (Estimated); Results first posted 2018-10-22 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-01

CONDITIONS: Failed Back Surgery Syndrome
MeSH Terms: conditions — Failed Back Surgery Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SQS plus OMM (Experimental): subcutaneous nerve stimulation plus optimized medical management
  Interventions: Device: subcutaneous nerve stimulation; Other: Optimized Medical Management
- OMM (Active Comparator): optimized medical management
  Interventions: Other: Optimized Medical Management

INTERVENTIONS:
Device: subcutaneous nerve stimulation — subcutaneous nerve stimulation plus optimized medical management
  Arms: SQS plus OMM
Other: Optimized Medical Management — Optimized medical management

SUMMARY:
The purpose of this study is to compare the effectiveness of peripheral nerve stimulation utilizing a subcutaneous lead implant technique (SQS) plus optimized medical management (OMM) versus OMM alone in patients suffering from back pain due to Failed Back Surgery Syndrome (FBSS).

ELIGIBILITY:
Inclusion Criteria:

1. Provides written Patient Informed Consent/Patient Information Sheet prior to study-related activities being conducted
2. ≥ 18 years of age at time of informed consent
3. Willing and available to attend visits as scheduled and to comply with the study protocol
4. Willing and able to undergo assessments as part of the evaluation for eligibility and endpoints
5. Willing and able to use the external neurostimulator, recharging equipment (if applicable), and patient programmer per the schedule required by the protocol
6. Diagnosed with FBSS (i.e.):

   * Has had persistent pain for 6 months following most recent anatomically correct, successful surgery AND
   * There are no further therapeutic surgical options available as assessed by appropriate investigation
7. Back pain is considered intractable and has been adequately treated (failed an appropriate trial of at least 3 different classes of back pain treatments (pharmaceutical and/or non-pharmaceutical))
8. Is an appropriate implant candidate for the SQS system

Exclusion Criteria:

1. Has been or is currently being treated with spinal cord stimulation, subcutaneous nerve stimulation, peripheral nerve stimulation or an implantable intrathecal drug delivery system
2. Evidence of an active disruptive psychiatric disorder that is significant enough to impact the perception of pain, compliance to intervention and/or ability to evaluate treatment outcome, as determined by the investigator
3. Has a pain condition unrelated to FBSS that is severe enough to overshadow the FBSS pain in the opinion of the investigator
4. Spinal instability or anatomic compression that requires further surgery
5. Spinal fusion at more than 3 vertebral levels
6. Currently enrolled in or plans to enroll in any concurrent drug and/or device study that may confound the results of this study
7. Allergic or has shown hypersensitivity to any materials of the device system which come in contact with the body
8. History of coagulation disorder or lupus erythematosus
9. Involved in current litigation regarding back pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2012-11; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sam Eldabe, MD, Principal Investigator — The James Cook Hospital
Locations (26):
- Australia (3):
  - Hunter Pain Clinic, Broadmeadow
  - Greenslopes Private Hospital, Greenslopes
  - Royal North Shore Hospital, St Leonards
- Austria (3):
  - Krankenhaus der Elisabethinen, Graz
  - Krankenhaus der Landes Kärnten, Klagenfurt
  - Krankenhaus der Barmherzigen Brüder, Vienna
- Belgium (4):
  - ZNA Middelheim, Antwerp
  - AZ Sint Jan, Bruges
  - INDC Jolimont, La Louvière
  - Pijnkliniek Stedelijk Ziekenhuis, Roeselare
- France (5):
  - Clinique Mutualiste de la porte de l'Orient, Lorient
  - Hospices civils de LYON, Lyon
  - Clinique Brétéché, Nantes
  - Fondation Rothschild, Paris
  - Hopital Purpan, Toulouse
- Germany (3):
  - Universitätsklinikum Köln, Cologne
  - Märkische Kliniken GmbH / Marienhospital Letmathe, Iserlohn-Letmathe
  - Universitätsklinikum Jena, Jena
- Tel Aviv Medical Center, Tel Aviv, Israel
- Netherlands (4):
  - Rijnland Ziekenhuis, Alphen aan den Rijn
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Amphia Ziekenhuis, Oosterhout-Breda
  - Maasstad Ziekenhuis, Rotterdam
- Hospital Universitario del Rio Hortega, Valladolid, Spain
- Hopital de Morges, Morges, Switzerland
- The James Cook Hospital, Middlesbrough, United Kingdom

REFERENCES:
- [Derived] Eldabe S, Kern M, Peul W, Green C, Winterfeldt K, Taylor RS. Assessing the effectiveness and cost effectiveness of subcutaneous nerve stimulation in patients with predominant back pain due to failed back surgery syndrome (SubQStim study): study protocol for a multicenter randomized controlled trial. Trials. 2013 Jun 25;14:189. doi: 10.1186/1745-6215-14-189. PMID 23799929

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject enrolled in the study on January 11, 2013. The last subject was enrolled on January 15, 2016 and all subject visits were stopped as of the study termination date of February 12, 2016.
Pre-assignment Details: Patients were considered enrolled in the study upon signing an Informed Consent Form. Enrolled subjects then completed additional assessments and were provided a diary to record ther back and leg pain intensity. Upon completion of the at-home diary, eligibility was reassessed based on pain scores. Eligible subjects were then randomized.
Groups:
- SQS+OMM: Subcutaneous nerve stimulation (SQS) plus optimized medical management (OMM)
- OMM Alone: Optimized Medical Management alone (OMM)
Period: Overall Study
Arm/Group | SQS+OMM | OMM Alone
Started | 56 | 60
Completed | 38 | 36
Not Completed | 18 | 24
Not completed — Early study termination | 10 | 14
Not completed — Withdrawal by Subject | 3 | 7
Not completed — Protocol Violation | 2 | 3
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SQS+OMM | OMM Alone | Total
Number analyzed (Participants) | 56 | 60 | 116
Age, Continuous [Mean (Standard Deviation); unit: years] — Mean age at time of enrollment (in years)
  years | 50.9 (10.9) | 52.2 (11.4) | 51.6 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Percentage of males and females
  Participants
    Female | 32 | 34 | 66
    Male | 24 | 26 | 50
Pain intensity at baseline [Mean (Standard Deviation); unit: units on a scale] — Pain intensity was measured by a 100 mm visual analog scale (VAS), with 0 representing no pain and 100 representing the worst pain imaginable.
  units on a scale
    Back pain | 68.8 (13.4) | 70.1 (14.0) | 69.5 (13.7)
    Leg pain | 8.9 (10.8) | 6.8 (11.5) | 7.8 (11.2)

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness of Treatment on Reduction of Back Pain Intensity
Description: Percentage of participants who responded to the treatment, where response was defined as ≥ 50% reduction in back pain intensity as measured by Visual Analog Scale from baseline to the 9-month follow-up visit. Pain intensity was measured by a 100 mm Visual Analog Scale, with 0 representing no pain and 100 representing the worst pain imaginable.
Time Frame: 9 months
Population: The Intent-to-Treat patient set (ITT) consists of all subjects as they were randomized into the study.
  The As Treated consists of all patients of the ITT patient set, but excludes those with major protocol deviations; they are analysed according to last treatment received before the actual assessment, without replacement of missing data.
Measure: Number (95% Confidence Interval); unit: Percentage of responders
Arm/Group | SQS+OMM | OMM Alone
Number analyzed (Participants) | 56 | 60
Percentage of responders
  Intent to treat | 33.9 [21.5 to 46.3] | 1.7 [0.0 to 4.9]
  As treated: number analyzed (Participants) | 30 | 35
  As treated | 56.7 [38.9 to 74.4] | 2.9 [0.0 to 8.4]
Statistical Analysis 1: Comparison: SQS+OMM vs OMM Alone; Subjects with missing information were considered in the test and computation of the proportion for ITT; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Nominal alpha of 4% was predefined for the final analysis

2. Secondary Outcome: Average Change in Back Pain Intensity
Description: Average change in back pain intensity from baseline to the 6 and 9-month follow-up visits. Pain intensity was measured by a 100 mm Visual Analog Scale, with 0 representing no pain and 100 representing the worst pain imaginable. A reduction in average pain score is indicated by a negative number.
Time Frame: 6 and 9 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SQS+OMM | OMM Alone
Number analyzed (Participants) | 56 | 60
units on a scale
  Intent to treat: Abs change in back pain at 6 mo | -33.7 (26.4) | -0.6 (14.3)
  Intent to treat: Abs change in back pain at 9 mo | -33.3 (24.5) | -2.7 (16.0)
  As treated: Absolute change in back pain at 6 mo: number analyzed (Participants) | 30 | 35
  As treated: Absolute change in back pain at 6 mo | -35.0 (25.5) | -2.9 (12.5)
  As treated:Absolute change in back pain at 9 mo: number analyzed (Participants) | 30 | 35
  As treated:Absolute change in back pain at 9 mo | -35.9 (25.3) | -4.1 (14.8)
Statistical Analysis 1: Comparison: SQS+OMM vs OMM Alone; Test type: Superiority or Other; p < 0.0001, Regression, Linear — Nominal alpha of 5% was pre-defined for the final analysis

3. Secondary Outcome: Back Pain Responder Rate (≥50%) at 6 Months
Description: Percentage of participants who responded to the treatment, where response was defined as ≥ 50% reduction in back pain intensity as measured by Visual Analog Scale from baseline to the 6-month follow-up visit. Pain intensity was measured by a 100 mm Visual Analog Scale, with 0 representing no pain and 100 representing the worst pain imaginable.
Time Frame: 6 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of responders
Arm/Group | SQS+OMM | OMM Alone
Number analyzed (Participants) | 56 | 60
Percentage of responders
  Intent to treat | 26.8 [15.2 to 38.4] | 1.7 [0.0 to 4.9]
  As treated: number analyzed (Participants) | 30 | 35
  As treated | 40.0 [22.5 to 57.5] | 2.9 [0.0 to 8.4]
Statistical Analysis 1: Comparison: SQS+OMM vs OMM Alone; Subjects with missing information were considered in the test and computation for ITT; Test type: Superiority or Other; p = 0.0002, Fisher Exact — Nominal alpha of 5% was pre-defined for the final analysis

4. Secondary Outcome: Back Pain Responder Rate (≥30%) at 9 Months
Description: Percentage of participants who responded to the treatment, where response was defined as ≥ 30% reduction in back pain intensity as measured by Visual Analog Scale from baseline to the 9-month follow-up visit. Pain intensity was measured by a 100 mm Visual Analog Scale, with 0 representing no pain and 100 representing the worst pain imaginable.
Time Frame: 9 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of responders
Arm/Group | SQS+OMM | OMM Alone
Number analyzed (Participants) | 56 | 60
Percentage of responders
  Intent to treat | 44.6 [31.6 to 57.7] | 5.0 [0.0 to 10.5]
  As treated: number analyzed (Participants) | 30 | 35
  As treated | 70.0 [53.6 to 86.4] | 11.4 [0.9 to 22.0]
Statistical Analysis 1: Comparison: SQS+OMM vs OMM Alone; Subjects with missing information were considered in the test and computation for ITT; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Nominal alpha of 5% was pre-defined for the final analysis

ADVERSE EVENTS:
Time Frame: Adverse events were collected from randomization through the study end (up to 36 months follow-up).
Description: All adverse event were collected, regardless of relationship to device or therapy. Whether an event met the criteria of serious was determined by the study site. The Safety Patient Set was pre-defined as all subjects of the Intent to Treat patient set (n=116) who started any of the study procedures, independent of the treatment they had been randomized to. There were 115 patients included in the Safety Patient Set: 55 patients in the SQS+OMM and 60 patients in the OMM alone arm.
Arm/Group | SQS+OMM | OMM Alone
Serious Adverse Events (participants affected / at risk) | 19/55 | 9/60
Other Adverse Events (participants affected / at risk) | 18/55 | 17/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SQS+OMM (N=55) | OMM Alone (N=60)
Cardiac disorder (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Diaphragmatic hernia (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Device stimulation issue (General disorders) | 2 | 0
Drug withdrawal syndrome (General disorders) | 1 | 1
Implant site paraesthesia (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Therapeutic product ineffective (General disorders) | 2 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Implant site infection (Infections and infestations) | 2 | 0
Skin infection (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
C-reactive protein abnormal (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Muscle contractions involuntary (Nervous system disorders) | 1 | 0
Mental disorder (Psychiatric disorders) | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Drug detoxification (Surgical and medical procedures) | 0 | 1
Haemorrhoid operation (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SQS+OMM (N=55) | OMM Alone (N=60)
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Food poisoning (Gastrointestinal disorders) | 0 | 1
Gastric polyps (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Oral lichen planus (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Adverse drug reaction (General disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Device stimulation issue (General disorders) | 1 | 0
Drug withdrawal syndrome (General disorders) | 2 | 2
Fatigue (General disorders) | 0 | 3
Hernia (General disorders) | 0 | 1
Implant site pain (General disorders) | 3 | 1
Swelling (General disorders) | 0 | 1
Temperature intolerance (General disorders) | 1 | 0
Therapeutic product ineffective (General disorders) | 1 | 0
Liver injury (Hepatobiliary disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Breast infection (Infections and infestations) | 0 | 1
Candidiasis (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Implant site infection (Infections and infestations) | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Incision site pain (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Splinter (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 2
Blood cholesterol increased (Investigations) | 0 | 1
Blood pressure difference of extremities (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1
Cardiac murmur (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0
Serum ferritin increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 2
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 2
Dizziness (Nervous system disorders) | 1 | 1
Drop attacks (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 2
Migraine (Nervous system disorders) | 0 | 1
Myelopathy (Nervous system disorders) | 1 | 0
Myoclonus (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Sedation (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Thoracic outlet syndrome (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Nightmare (Psychiatric disorders) | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 1
Genital haemorrhage (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash follicular (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hot flush (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study Publication Committee manages and oversees publications generated from the study. The sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor can require changes to the communication related to patentable and copyrightable material and can extend the embargo.